CLINICAL TRIAL: NCT05051358
Title: Therapeutic Endoscopic Ultrasound for Gastrointestinal Disorders: A Multicenter Registry
Brief Title: Therapeutic Endoscopic Ultrasound for Gastrointestinal Disorders: A Multicenter Registry Study
Acronym: TEUS Registry
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Advanced Endoscopy Research, Robert Wood Johnson Medical School Rutgers University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro2020002795
Record Dates: First submitted 2021-09-03; First posted 2021-09-21 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Therapeutic Endoscopic Ultrasound; Advanced Endoscopy; Therapeutic Endoscopy; Interventional Endoscopy; Interventional Endoscopic Ultrasound; Gastro-Intestinal Disorder; Gastrointestinal Disease; Gastrointestinal Cancer; Gastrointestinal Dysfunction; Gastrointestinal Fistula; Gastrointestinal Infection; Gastrointestinal Injury; Pancreatic Disease; Bile Duct Diseases
MeSH Terms: conditions — Digestive System Diseases; Gastrointestinal Diseases; Gastrointestinal Neoplasms; Digestive System Fistula; Pancreatic Diseases; Bile Duct Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects undergoing Therapeutic Endoscopic Ultrasound: Procedures that will be captured include:
  EUS- ERCP, Endoscopic Hepatology - EUS, EUS-Coils placement, EUS Glue injection, EUS-Fiducial placement, EUS-Neurolysis, EUS-Stent placement, EUS-alcohol injection, EUS-guided Ablation, EUS-guided anastomosis, EUS Guided ERCP for gallbladder, pancreatic duct or biliary duct drainage, EUS guided - Hemostasis, EUS guided- Therapy for cancer or premalignant lesion (Injection, neurolysis, fiducial, aspiration, RFA ), EUS - Fluid Collection, abscess or cavity drainage, EUS - Guided Ductal Drainage, EUS - Guided Anastomosis
  Interventions: Procedure: Therapeutic Endoscopic Ultrasound

INTERVENTIONS:
Procedure: Therapeutic Endoscopic Ultrasound — Therapeutic Endoscopic Ultrasound or Interventional Endoscopy for Gastrointestinal Indications

SUMMARY:
The purpose of this retrospective chart-review registry study is to evaluate the safety profile, efficacy profile and cost-effectiveness of the various therapeutic endoscopic ultrasound (EUS) procedures (for benign and malignant gastrointestinal disorders).

1. To assess the clinical and technical success rates of EUS-Guided interventions
2. To document the impact of therapeutic EUS procedures on the management of gastrointestinal disorders including malignancies through cost effective analyses.
3. Compare endoscopic interventions to non-endoscopic interventions for the same clinical indications and evaluate safety and efficacy.

DETAILED DESCRIPTION:
Our tertiary-care institution performs clinically-indicated therapeutic Endoscopic Ultrasound (TEUS) guided interventions, including biliary and pancreatic drainage, for both malignant and benign gastrointestinal indications in more than 2000 patients annually.

Procedures such as biliary and/or pancreatic sphincterotomy, stents placement (metallic or plastic) and removal for revision, cysts and pseudocysts drainage are conducted in patients suffering from pancreatico-biliary disorders, gastrointestinal disorders and esophageal disorders.

TEUS procedures are less invasive approach than surgery. Moreover, they can be available to patients who are ineligible for surgery or who have refused more aggressive surgical intervention.

They improve quality of life and extend survival duration.

Currently, there is limited multi-center data on therapeutic endoscopy clinical outcomes and standardized treatment algorithms in western populations. Due to continuing variations in therapeutic EUS procedures, as well as introduction of some TEUS procedure accessories; it is necessary to periodically evaluate the efficacy and safety of specific TEUS procedures and accessories for several indications to check for improved clinical outcomes.

Evaluation of these clinical details would help us compare them to conventional treatment modalities within our current facility and scope of practice; and consequently, help us identify safe and cost-effective treatment techniques, develop treatment algorithms and improve clinical management of patients at RWJMS and other tertiary-care centers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing Interventional Therapeutic Endoscopic Ultrasound Procedures for Gastrointestinal indications

Exclusion Criteria:

* Subjects not undergoing Interventional Therapeutic Endoscopic Ultrasound Procedures for Gastrointestinal indications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects undergoing Interventional Therapeutic Endoscopic Ultrasound Procedures for Gastrointestinal indications
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-02-11 (Actual); Primary Completion 2023-12-10 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Procedure | Upto 2 years
  Technical and clinical success rates
Safety of procedure | Upto 2 years
  Type, frequency and intensity of adverse events

SECONDARY OUTCOMES:
Cost Effectiveness | Upto 2 years
  Total cost associated with procedures

CONTACTS AND LOCATIONS:
Overall Officials: Michel Kahaleh, MD, Principal Investigator — Advanced Endoscopy Research, Robert Wood Johnson Medical School Rutgers University
Locations (1):
- Advanced Endoscopy Research, Robert Wood Johnson Medical School Rutgers University, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be made available to other out-of-site researchers

REFERENCES:
- [Derived] Karanfilian B, Tyberg A, Sarkar A, Shahid HM, Simon A, Reinoso K, Bapaye A, Gandhi A, Gadhikar HP, Dorwat S, Raina H, Ansari J, Nieto J, Qadir N, Porfilio MG, Arevalo-Mora M, Puga-Tejada M, Alcivar-Vasquez J, Robles-Medranda C, Ardengh JC, Bareket R, Liao K, Patel R, Pimpinelli S, Gaidhane M, Kahaleh M. Impact of COVID-19 Infection on Pancreato-Biliary Diseases Requiring Endoscopic Retrograde Cholangiopancreatography. Dig Dis Sci. 2024 Aug;69(8):3015-3018. doi: 10.1007/s10620-024-08454-1. Epub 2024 May 7. PMID 38713274
- [Derived] Tyberg A, Duarte-Chavez R, Shahid HM, Sarkar A, Simon A, Shah-Khan SM, Gaidhane M, Mohammad TF, Nosher J, Wise SS, Needham V, Kheng M, Lajin M, Sojitra B, Wey B, Dorwat S, Raina H, Ansari J, Gandhi A, Bapaye A, Shah-Khan SM, Krafft MR, Thakkar S, Singh S, Bane JR, Nasr JY, Lee DP, Kedia P, Arevalo-Mora M, Del Valle RS, Robles-Medranda C, Puga-Tejada M, Vanella G, Ardengh JC, Bilal M, Giuseppe D, Arcidiacono PG, Kahaleh M. Endoscopic Ultrasound-Guided Gallbladder Drainage Versus Percutaneous Drainage in Patients With Acute Cholecystitis Undergoing Elective Cholecystectomy. Clin Transl Gastroenterol. 2023 Jun 1;14(6):e00593. doi: 10.14309/ctg.0000000000000593. PMID 37141073
- [Derived] Tyberg A, Sarkar A, Shahid HM, Shah-Khan SM, Gaidhane M, Simon A, Eisenberg IA, Lajin M, Karagyozov P, Liao K, Patel R, Zhao E, Martinez MG, Artifon EL, Lino AD, Vanella G, Arcidiacono PG, Kahaleh M. EUS-Guided Biliary Drainage Versus ERCP in Malignant Biliary Obstruction Before Hepatobiliary Surgery: An International Multicenter Comparative Study. J Clin Gastroenterol. 2023 Oct 1;57(9):962-966. doi: 10.1097/MCG.0000000000001795. PMID 36730114